CLINICAL TRIAL: NCT00880347
Title: Blood Gene Expression Signature in Patients Diagnosed With Probable Alzheimer's Disease Compared to Patients Suffering From Other Types of Dementia : A Prospective Study for a Blood Diagnostic Test in Alzheimer's Disease - (Protocol n° EHTAD/002).
Brief Title: Blood Gene Expression Signature in Patients Diagnosed With Probable Alzheimer's Disease Compared to Patients Suffering From Other Types of Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Exonhit (Industry)
Responsible Party: Professor Bruno Vellas, MD, University of Toulouse - Purpan - Casselardit Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: EHTAD/002
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer's disease; Other dementia; Vascular dementia; Mixed dementia; Parkinson's Disease dementia; Lewy bodies dementia; Frontotemporal dementia; Blood signature; Diagnosis; SpliceArray (tm); Alzheimer's Disease and other non-AD dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia; Dementia, Vascular; Mixed Dementias; Lewy Body Disease; Frontotemporal Dementia; Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alzheimer's Disease (Other): Group of patients clinically diagnosed with probable AD
  Interventions: Device: Blood sampling
- Non-AD dementia (Other): Group of patients clinically diagnosed with one of the 5 most frequent non-AD dementia : vascular dementia, mixed dementia, frontotemporal dementia, Lewy bodies dementia, Parkinson's disease dementia.
  Interventions: Device: Blood sampling
- control subjects (Other): Group of control subjects without any clinical cognitive impairment.
  Interventions: Device: Blood sampling

INTERVENTIONS:
Device: Blood sampling — Venous blood sampling in PaxGene tubes intended to collect blood RNA that will be then analyzed using SpliceArray (tm) technology for transcriptomic profile. sAPPalpha levels will be also dosed. Clinical data to be collected in parallel (medical history, concomitant treatment, MMSE,clinical examination,...)

SUMMARY:
The objective of the study is to define the performance of blood-based signatures for Alzheimer's Disease (AD) in different patients populations including AD, non-AD dementia, and non-demented controls.

DETAILED DESCRIPTION:
The main objective of the study is to define the performance of blood-based transcriptomic signatures for AD, identified using SpliceArray tm technology, in the intended use population of patients suffering from dementia, including AD and the most common non-AD dementia (Lewy Bodies dementia, vascular dementia, fronto-temporal dementia, dementia due to Parkinson's Disease, and mixed dementia). A group of non-demented subjects will serve as a control reference.

ELIGIBILITY:
Inclusion Criteria:

1. AD group :

   * Male or female patient, aged ≥ 40 years old included at entry.
   * Patients having a clinical diagnosis of probable AD according to DSM-IV TR [F00.xx] and National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
   * Written informed consent obtained from the patient or, if appropriate, from legal representative according to local laws and regulations.
   * Evidence that brain imaging (either cerebral CT-scan or cerebral MRI) was performed to settle the AD diagnosis, and that the results are compatible with AD diagnosis.
   * Neurological exam without any particularities or without any specific focal signs likely to be related to other conditions than AD.
   * Patient compliant with study procedures.
2. Non AD demented group :

   * Male or female patient, aged ≥ 40 years old included at entry.
   * Patients having a clinical diagnosis of dementia which can be one of the following :
   * VaD according to NINDS-AIREN criteria or,
   * LBD according to McKeith's criteria, or,
   * FTD according to Neary's or Lund & Manchester criteria or,
   * PDD according to DSM-IV TR criteria [F02.x] or,
   * Mixed dementia which is defined in this study as patients fulfilling DSM-IV TR criteria [F02.8] for dementia with multiple aetiologies focussing on dementia of Alzheimer type with secondary occurrence of vascular dementia.
   * Written informed consent obtained from the patient or, if appropriate, from legal representative according to local laws and regulations.
   * Evidence that brain imaging (either cerebral CT-scan or cerebral MRI) was performed to settle the diagnosis of dementia, and that the results are compatible with the diagnosis of dementia.
   * Absence of other signs or symptoms that may be better related to another type of dementia than the current dementia diagnosis.
   * Patient compliant with study procedures.
3. Cognitive impairment-free control group :

   * Male or female subject, aged ≥ 60 years old included at entry.
   * Written informed consent obtained from the subject.
   * Absence of spontaneously reported significant cognitive complaints from the subject at entry.
   * MMSE ≥ 27 at entry.
   * Subject with no impairment in daily living activities.
   * Subject compliant with study procedures.

Exclusion Criteria:

1. AD group :

   * Any pathology, medical condition or symptoms that may lead to reconsider the initial diagnosis of probable AD, or that may rend the initial diagnosis of probable AD doubtful at entry, according to the opinion of the investigator.
   * Current or recent history of drug or alcohol abuse or dependence.
   * Diagnostic of Mild Cognitive Impairment defined by subjective complaints from the patient regarding memory and/or cognitive symptoms, objective memory and/or cognitive impairment at testing but not meeting AD diagnostic criteria, and not affecting daily living activities.
   * Current diagnosis of brain tumour.
   * Any current pathology or medical condition, for which blood sampling may involve a risk for the patient's health, according to the opinion of the investigator.
   * Pregnancy.
   * Patient who is not registered at "Sécurité Sociale".
   * Current participation in another study using an investigational non-marketed product.
2. Non-AD demented group :

   * Any pathology, medical condition or symptoms that may lead to reconsider the initial diagnosis of dementia the patient is suffering from, or that may rend the initial diagnosis of dementia doubtful at entry, according to the opinion of the investigator.
   * Diagnostic of Mild Cognitive Impairment defined by subjective complaints from the patient regarding memory and/or cognitive symptoms, objective memory and/or cognitive impairment at testing but not meeting the diagnostic criteria for dementia, and not affecting daily living activities.
   * Current diagnosis of brain tumour.
   * Any current pathology or medical condition for which blood sampling may involve a risk for the patient's health, according to the opinion of the investigator.
   * Current or recent history of drug or alcohol abuse or dependence.
   * Pregnancy.
   * Patient who is not registered at "Sécurité Sociale".
   * Current participation in another study using an investigational non-marketed product.
3. Cognitive impairment-free control group :

   * Subject spontaneously complaining from significant cognitive impairment.
   * Known family history of dementia.
   * Diagnosis of any type of dementia (either AD or non-AD dementia), Mild Cognitive Impairment, or any current or past history of CNS pathology (including but not limited to brain injury, brain tumour, stroke, normal pressure hydrocephalus, Parkinson's disease, epilepsy, multiple sclerosis,…) that may be responsible for the occurrence of dementia.
   * History or current clinically significant psychiatric pathology (including but not limited to psychotic disorders, bipolar disorder, personality disorders).
   * Current major depressive disorder, either treated or not, associated with clinically significant symptoms.
   * Any current pathology or medical condition for which blood sampling may involve a risk for the subject's health, according to the opinion of the investigator.
   * Current or recent history (within one month) of clinically significant pathology, medical condition (including hospitalization) or symptoms. However, chronic diseases or medical conditions which are considered stable are accepted, provided that they are compatible with other study selection criteria.
   * Current or recent history of drug or alcohol abuse or dependence.
   * Subject who is not registered at "Sécurité Sociale".
   * Current participation in another study using an investigational non-marketed product.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To define the test performance of the blood expression signatures in the intended use population of demented patients to differentiate AD patients from non-AD demented patients. | day 1 (cross-sectional study)

SECONDARY OUTCOMES:
Performance of blood signatures (AD versus control, AD vs each individual type of non-AD dementia,...). Specificity of the blood signatures versus NINCDS-ADRDA criteria. Exploratory assessment of clinical parameters that may influence blood signature. | day1 (cross-sectional study)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier SOL, MD, Study Director — Exonhit; Bruno Vellas, MD, Principal Investigator — Purpan- Casselardit Hospital - Toulouse University
Locations (21):
- France (21):
  - Hôpital Privé Les Magnolias, Ballainvilliers
  - Cabinet Médical, Bergerac
  - Centre Médical, Dijon
  - Cabinet Médical, La Seyne-sur-Mer
  - Cabinet Médical, Le Vésinet
  - Clinique Léopold Bellan, Magnanville
  - Cabinet Médical, Marseille
  - Centre Médical, Montpellier
  - Cabinet Médical, Montpellier
  - CMRR Gui de Chauliac Hospital, Montpellier
  - CHU Nantes Hôpital Laennec, Nantes
  - ClinOuest network, Nantes
  - Cabinet Médical 2, Nice
  - Cabinet Médical, Nice
  - Cabinet Médical, Paris
  - Centre Médical, Rambouillet
  - Cabinet Médical, Rodez
  - Cabinet Médical, Rueil-Malmaison
  - Cabinet Médical, Saint-Brieuc
  - Purpan-Casselardit Hospital - University of Toulouse, Toulouse
  - CDPRV Le Capitole, Valence